CLINICAL TRIAL: NCT03092167
Title: Physical Training in Patients With Idiopathic Inflammatory Myopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Samuel Katsuyuki Shinjo, PhD, Principal Investigator, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MYO-HCFMUSP-02
Record Dates: First submitted 2017-03-09; First posted 2017-03-27 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Idiopathic Inflammatory Myopathies; Physical Activity
MeSH Terms: conditions — Myositis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 15 idiopathic inflammatory myopathies submmited to physical exercises 15 idiopathic inflammatory myopathies not submmited to physcial exercises 10 healthy individuals
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Case (Active Comparator): Patients: this group will be submitted to 12-weeks, twice/week, physical exercises.
  Interventions: Other: Physical exercises
- Control (No Intervention): Patients: this group will not be submitted to 12-weeks, twice/week, physical exercises.
- Healthy control (No Intervention): Volunteers: this group will not be submitted to 12-weeks, twice/week, physical exercises.

INTERVENTIONS:
Other: Physical exercises — Physical exercises
  Arms: Case

SUMMARY:
Physical training may improve physical capacity and health parameters in various systemic autoimmune diseases, including idiopathic inflammatory myopathies. Therefore, the present study will assess the role of an exercise training program in patients with idiopathic inflammatory myopathies.

DETAILED DESCRIPTION:
To assess the impact of 12-weeks of physical training in patients with idiopathic inflammatory myopathies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DM / PM according to the criteria of Bohan and Peter (1975)
* Both genders and age ≥ 18 years
* Use of prednisone ≤ 0.5 mg/kg/day in the last three months. The dose of prednisone will be kept fixed throughout the study
* Physically inactive

Exclusion Criteria:

* Disease relapsing
* Neoplasia associated-myositis
* Overlapping myositis
* Use of lipid-lowering drugs
* Smoking
* Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary test | 12 weeks
  Patients will undertake a maximal graded exercise test on a treadmill, with increments in velocity and grade at every minute until volitional exhaustion. VO2peak will be considered as the average of the final 30 s of the test. Ventilatory threshold (VAT) will be determined when ventilatory equivalent for VO2 (VE/VO2) increased without a concomitant increase in ventilatory equivalent for carbon dioxide (VE/VCO2). Respiratory compensation point (RCP) will be determined when VE/VO2 and VE/VCO2 increased simultaneously.

SECONDARY OUTCOMES:
Serum cytokines | 12 weeks
  Blood samples will be centrifuged at 3000 rpm for 15 min at 4°C, and the serum aliquot will be stored at -80°C for subsequent analyses. Cytokines (i.e., IL-6, TNF alpha, IFN gamma) will be measured using a multiplex human panel (Milliplex Map, Millipore, Billerica, MA, USA). Data analysis will be performed through Luminex xMAP Technology, according to the manufacturer's instructions.
Strength muscle tests | 12 weeks
  The dynamic 1-RM for the leg-press and the bench-press exercises, arm curl (with the dominant arm).
Muscle biopsies | 12 weeks
  After local anesthesia, a cutaneous incision will be made in lateral thigh face. The biopsy will be done using the Bergstrom needle. Histological (hematoxylin and eosin)/immunohistochemical (CD4, CD8, CD68, CD20, C5b-9, MHCI, MHCII, CD31) analysis will be performed in muscle samples (at baseline and after 12 weeks) in all patients (present study)
Functional muscle tests | 12 weeks
  Isometric strength (assessed by handgrip, with the dominant arm) will be assessed at baseline and after the intervention. Muscle function will be evaluated through the TUG and the TST tests.
Myositis Disease Activity Assessment Tool | 12 weeks
  This partially validated tool measures the degree of disease activity of extra-muscular organ systems and muscle. This is a combined tool that includes the Myositis Disease Activity Assessment Visual Analogue Scales (MYOACT), which is a series of physician's assessments of disease activity, and the Myositis Intention to Treat Activity Index (MITAX).
Muscle enzymes | 12 weeks
  This partially validated tool measures the serum activities of at least 2 of the 4 muscle-associated enzymes including creatine phosphokinase (CK), the transaminases (ALT, AST), lactate dehydrogenase (LD) and aldolase.
Health Assessment Questionnaire | 12 weeks
  Especific questionnaire (health assessment questionnaire). Pontuaction 0.00-3.00
Manual Muscle Testing | 12 weeks
  This partially validated tool assesses muscle strength using manual muscle testing (MMT). A 0 - 10 point scale is proposed for use. An abbreviated group of 8 proximal, distal, and axial muscles performs similarly to a total of 24 muscle groups, and is also proposed for use for research studies.
Patient/Parent Global Activity | 12 weeks
  This partially validated tool measures the global evaluation by the patient, or by the parent if the patient is a minor, of the patient's overall disease activity at the time of assessment using a 10 cm. visual analogue scale.
Physician Global Activity | 12 weeks
  This partially validated tool measures the global evaluation by the treating physician of the overall disease activity of the patient at the time of assessment using a 10 cm. visual analogue scale and a 5 point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel K Shinjo, PhD, Principal Investigator — Universidade de Sao Paulo - Rheumatology Division
Locations (1):
- Samuel Katsuyuki Shinjo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borges IBP, de Oliveira DS, Marie SKN, Lenario AM, Oba-Shinjo SM, Shinjo SK. Exercise Training Attenuates Ubiquitin-Proteasome Pathway and Increases the Genes Related to Autophagy on the Skeletal Muscle of Patients With Inflammatory Myopathies. J Clin Rheumatol. 2021 Sep 1;27(6S):S224-S231. doi: 10.1097/RHU.0000000000001721. PMID 34227790